CLINICAL TRIAL: NCT06344611
Title: Incidence & Predictive Factors of Recompensation in Children With Decompensated Cirrhosis as Per the Baveno VII Criteria
Status: Not yet recruiting | Type: Observational
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Other Study IDs: ILBS-DCLD-01
Record Dates: First submitted 2024-03-27; First posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-03

CONDITIONS: Decompensated Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Decompensated Cirrhosis
  Interventions: Other: Other

INTERVENTIONS:
Other: Other — It is an observational study. Subjects will receive the treatment as per institute protocol.

SUMMARY:
Cirrhosis is a leading cause of morbidity and mortality world- wide and can develop on the basis of repetitive and/or chronic liver injury due to toxic, infectious, metabolic and genetic pathogenic factors. Traditionally, the natural history of cirrhosis has often been considered a one-way street, with a definite and irreversible progression from a compensated to a decompensated disease stage. But recent data has shown that if the underlying etiology can be successfully treated, cirrhosis can regress and recompensation of liver disease can occur. Hence, in this study we want to evaluate the incidence and predictive factors of recompensation in pediatric subjects with decompensated cirrhosis as per the Baveno VII criteria. We would also evaluate the predictive factors of recompensation in pediatric decompensated chronic liver disase (DCLD) subjects and would explore systemic and intestinal inflammatory markers as possible biomarkers for predicting recompensation in pediatric subjects with decompensated cirrhosis.

DETAILED DESCRIPTION:
Aim- To evaluate the incidence and predictive factors of recompensation in pediatric subjects with decompensated cirrhosis as per the Baveno VII criteria Primary objective: To determine the incidence of recompensation in pediatric subjects with decompensated cirrhosis as per Baveno VII criteria

Secondary objectives:

1. To evaluate the predictive factors of recompensation in pediatric DCLD subjects
2. To investigate the systemic and intestinal inflammatory markers as possible biomarkers for predicting recompensation in pediatric subjects with decompensated cirrhosis
3. To assess incidence of re-decompensation in patients with recompensation Study design: Prospective, Observational study. Study period:2 years (Aug 2023-Jul2025). Sample size: Time bound; All decompensated cirrhosis cases presenting to the institute during the study period will be included in the study.

Intervention: None, since it is an observational study only

* Monitoring and assessment:
* Along with standard tratment plan/investigatios (as per etiology), Liver function test, INR and Ultrasound abdomen would be done at 3 monthly interval.
* At baseline: Markers of Systemic Inflammation (serum levels of IL-6, TNFα, IL-1β; Monocyte/Basophil Frequency, NLR; CRP, Procalcitonin) and Intestinal Inflammation (Stool cytokines- IL-6, TNFα, IL-1β, IL-10)

ELIGIBILITY:
Inclusion Criteria:

1. < 18 years of age at presentation
2. Decompensated cirrhosis at baseline

   1. Cirrhosis:defined asliver histology findings (> F4 fibrosis as per Ishak system), and/or
   2. radiological findings of an irregular nodular liver with/out left/caudate liver enlargement
   3. Decompensation:defined as presence of ascites (any grade), and/orHE (overt), and/or variceal haemorrhage (endoscopy proven)
3. Fulfilling Recompensation criteria as per Baveno VII (2022) after treatment initiation
4. Sustained cure, suppression or removal of the underlying aetiology of cirrhosis

   a. Includes treatable etiologies like Hepatitis B, Autoimmune liver disease, Wilson disease, Budd Chiari syndrome, MLDs (like Galactosemia, Tyrosinemia, Bile acid synthetic defects)
5. Resolution of ascites and hepatic encephalopathy (HE) after discontinuation of diuretics and prophylactic therapies, as well as the absence of variceal bleeding for 12 months.
6. Sustained improvement of biochemical liver function, as as- sessed by serum albumin, bilirubin and INR (international normalized ratio) a. improvement in liver function parameters to values within normal ranges (albumin >35 g/L & INR < 1.5 & bilirubin < 2 mg/dl)

Exclusion Criteria:

1. refused consent
2. patients with liver cancer or other active malignancy
3. Any significant extrahepatic disease

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subjects visiting to ILBS with decompensated Chronic liver disease from Aug 2023 till April 2025.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-04-07 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
To determine the incidence of recompensation in pediatric subjects with decompensated cirrhosis as per Baveno VII criteria | 1.5 years

SECONDARY OUTCOMES:
To evaluate the predictive factors of recompensation in pediatric DCLD subjects | 1.5 years
To investigate the systemic and intestinal inflammatory markers as possible biomarkers for predicting recompensation in in pediatric subjects with decompensated cirrhosis. | 1.5 years
To assess incidence of re-decompensation in patients with recompensation. | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided